CLINICAL TRIAL: NCT07066735
Title: Comparison of the Efficacy and Safety of Combined Extracorporeal Shock- Wave Therapy (ESWT) With Phytotherapy Versus Each of Them Alone in Chronic Prostatitis Category ⅢB
Brief Title: Extracorporeal Shock-Wave Therapy (ESWT) vs Phytotherapy vs Combined in Treatment of Chronic Prostatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Younan Ramsis, Lecturer of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU RSS/2025
Record Dates: First submitted 2025-06-28; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Prostatitis (CP)
Keywords: Chronic prostatitis; ESWT; Phytotherapy; LUTS
MeSH Terms: interventions — saw palmetto extract; pygeum extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A ESWT and Phytotherapy (Experimental): First group will undergo ( ESWT -Transperineal- once a week for 8 consecutive weeks with a protocol of 3000 pulses each; pressure: 1.8-2.0 bar and a frequency of 10 Hertz (Hz) (Zhang et al . 2018) combined with Phytotherapy that contains powder extract of (saw palmetto , tomato , uva ursi , pygeum , pumpkin ) 1capsule twice daily.
  Interventions: Device: ESWT; Drug: Phytotherapy that contains powder extract of (saw palmetto , tomato , uva ursi , pygeum and pumpkin
- Group B: ESWT alone (Experimental): Transperineal- once a week for 8 consecutive weeks with a protocol of 3000 pulses each; pressure: 1.8-2.0 bar and a frequency of 10 Hertz (Hz)
  Interventions: Device: ESWT
- Group 3: Phytotherapy alone (Active Comparator): Phytotherapy that contains powder extract of (saw palmetto , tomato , uva ursi , pygeum , pumpkin ) 1capsule twice daily
  Interventions: Drug: Phytotherapy that contains powder extract of (saw palmetto , tomato , uva ursi , pygeum and pumpkin

INTERVENTIONS:
Device: ESWT — Transperineal Shockwaves that are applied once a week for 8 consecutive weeks with a protocol of 3000 pulses each; pressure: 1.8-2.0 bar and a frequency of 10 Hertz (Hz)
  Arms: Group A ESWT and Phytotherapy; Group B: ESWT alone
Drug: Phytotherapy that contains powder extract of (saw palmetto , tomato , uva ursi , pygeum and pumpkin — 1capsule tob be taken twice daily for one month.
  Arms: Group 3: Phytotherapy alone; Group A ESWT and Phytotherapy

SUMMARY:
to compare the efficacy and safety of ESWT combined with phytotherapy, ESWT alone and phytotherapy alone in treatment of chronic prostatitis.

DETAILED DESCRIPTION:
In this study the investigators will conduct a Prospective randomized clinical trial, patients will be randomized to 3 groups where they will use use radial waves device (INTELECT RPW SHOCKWAVE) By Chattanooga for ESWT. Another group will receive Phytothyrapy that will be capsules containing powder extract of saw palmetto , tomato , uvaursi , pygeum and pumpkin. while the last group will receive both.

ELIGIBILITY:
Inclusion Criteria:

* Perineal or pelvic pain or discomfort of at least 3 months
* NIH-CPSI total score greater than 15,
* Negative semen cultures for bacteria.

Exclusion Criteria:

* Evidence of bacteria in seminal culture tests,
* Urinary stones,
* Uncontrolled coagulopathy,
* Chronic bacterial prostatitis,
* Bladder and prostate cancer,
* Medications that could affect lower urinary tract function during the last month
* Serum prostate-specific antigen levels (PSA) more than 4 ng/mL
* History of prostate surgery or radiotherapy
* Perineal anatomical abnormalities
* Neurological abnormalities.
* Previous extensive pelvic injuries

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
compare the degree of symptoms relief between the three groups | pre intervenon, at 4 and 8 weeks post intervention and at 2 and 4 months post intervention.
  using National Institutes of Health-developed Chronic Prostatitis Symptom Index (NIHCPSI) that will be filled by the patients pre and post intervention at 4 weeks and 8 weeks, 2 and 4 months. It comprises three key domains: pain (scored from 0 to 21), urinary symptoms (0 to 10), and the impact on quality of life (0 to 12), with a total score range spanning from 0 to 43. Higher scores reflect more severe symptoms and a worse overall outcome, while lower scores indicate milder symptoms and a better clinical picture. Severity is typically interpreted as mild (0-9), moderate (10-18), severe (19-31), and very severe (32-43), making the scale valuable for both diagnosis and monitoring treatment progress.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Y. Yassin, Professor, Study Chair — Ain Shams University
Locations (1):
- AinShams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagenlehner FM, van Till JW, Magri V, Perletti G, Houbiers JG, Weidner W, Nickel JC. National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) symptom evaluation in multinational cohorts of patients with chronic prostatitis/chronic pelvic pain syndrome. Eur Urol. 2013 May;63(5):953-9. doi: 10.1016/j.eururo.2012.10.042. Epub 2012 Nov 2. PMID 23141933
- [Background] Sakr AM, Fawzi AM, Kamel M, Ali MM. Outcomes and clinical predictors of extracorporeal shock wave therapy in the treatment of chronic prostatitis/chronic pelvic pain syndrome: a prospective randomized double-blind placebo-controlled clinical trial. Prostate Cancer Prostatic Dis. 2022 Mar;25(1):93-99. doi: 10.1038/s41391-021-00464-8. Epub 2021 Oct 11. PMID 34635804
- [Background] Palmieri A, Cai T, Di Luise L, D'Alterio C, La Cava G, Cirigliano L, Di Giovanni A, Gallelli L, Capece M. Extracorporeal shock wave therapy in association with bromelain and escin for the management of patients affected by chronic prostatitis/chronic pelvic pain syndrome. Biomed Rep. 2022 Nov 25;18(1):7. doi: 10.3892/br.2022.1589. eCollection 2023 Jan. PMID 36544851